CLINICAL TRIAL: NCT00853398
Title: A Prospective (Non)-Randomized Controlled Multicenter Clinical Study Of the Genesis ii Total Knee System in Minimally Invasive Total Knee Arthroplasty
Brief Title: MINIMALLY INVASIVE SURGERY in Total Knee Arthroplasty
Acronym: MIS GEN II
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The results obtained 1 year after surgery were clearly indicative of the outcome and the investigators decided to terminate follow-up at that point.
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: MIS_GEN_II_6112003
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: Primary Osteoarthritis of the knee.
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Wound Closure Techniques

ARMS (2):
- Minimal Invasive Surgery, (Experimental)
  Interventions: Procedure: surgical technique
- Standard Surgical Technique (Active Comparator)
  Interventions: Procedure: surgical technique

INTERVENTIONS:
Procedure: surgical technique

SUMMARY:
Overall study design:

A prospective, randomized, multi-center clinical studies comparing the minimal invasive and the standard surgical total knee replacement technique (control) using the Genesis II total knee system. The study will collect efficacy, safety and socio-economical data over 2 years. An additional 5 years follow-up interval is optional. The objectives (short-term follow-up) of the study are to:

1. Assess whether the improvement in Pain and Range of motion per Knee Society scoring system and VAS score.
2. Assess whether there are any differences between the surgical techniques as regards complication rate.
3. Assess whether the hospital stay and the rehabilitation time (Straight leg raise, Active/passive ROM) of the patients differs between the two techniques.
4. Assess the x-ray mechanical alignment between the two techniques.

Attempts will be made to assess whether the collected peri-operative data (including incision length, blood loss, wound appearance, hospital readmissions and operative time) differs between the two surgical techniques.

The primary objectives (mid-term follow-up) of the study are to:

1. Improvement in Pain and Function per Knee Society Scoring system
2. Number and Extent of Radiographic Lucencies >2mm
3. Revision and knee-related adverse events
4. Improvement in Quality-of-life via the VAS score

5 investigational sites will participate and enroll a total of approximately 250 patients over a 12 months period. Thus, each site will enroll 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* require primary uni- or bilateral total knee arthroplasty; available for 2 year follow up; provide informed consent; is in stable health for cardio-pulmonary conditions.

Exclusion Criteria:

* inefficient femoral or tibial bone stock; BMI >35; fixed flexion deformity >15 degrees; knee flexion of <90 degrees; varus/valgus deformity >20 degrees; active local infection; conditions that would compromise the 2 years follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pain and Range of Motion on the short term as efficacy measurements. Occurence of Adverse Events as safety measurements | 1 year

SECONDARY OUTCOMES:
Occurence of Adverse Events and Radiolucent lines > 2mm Range of motion on the mid term | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Department, University Hospital, Tübingen, Germany